CLINICAL TRIAL: NCT01111383
Title: A Single Arm 48-Week Follow-on Safety Study to the Core Study (A Multicentre, Multinational, Open-Label, Randomised, Parallel Group Clinical Trial of Tobrineb®/Actitob®/Bramitob® (Tobramycin Solution for Nebulisation, 300mg Twice Daily in 4mL Unit Dose Vials) Compared to TOBI® in the Treatment of Patients With Cystic Fibrosis and Chronic Infection With Pseudomonas Aeruginosa)
Brief Title: A Single Arm 48-Week Follow-on Safety Study to a Core Study Comparing the Efficacy and Tolerability of Tobrineb®/Actitob®/Bramitob® Versus TOBI®
Acronym: CT03Ext
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMA-0631-PR-0010 Extension
Record Dates: First submitted 2010-04-13; First posted 2010-04-27 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; P. aeruginosa; tobramycin
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: tobramycin — 300mg/4ml solution, via a nebuliser, over a 48-week period in a twice-daily regimen, with 6 "on" cycles of 4 weeks duration during the 48-week period.
  Other Names: Tobrineb®/Actitob®/Bramitob®

SUMMARY:
This is a 48-week extension study to CMA-0631-PR-0010 Core Study. Patients who have a positive culture for P. aeruginosa at visit 4 of the first 8-week core study period and/or if deemed appropriate by the Investigators will be able to be included in the 48-week follow-on period (Extension Study) to continue the treatment only with Bramitob® (tobramycin nebuliser solution, 300 mg twice daily in 4 mL unit dose vials).

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of Core Study
* At least 6 years of age
* Males and females

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
to assess safety profile in terms of incidence of adverse events/adverse drug reactions, frequency of cystic fibrosis exacerbations, audiometric test, laboratory parameters (hematology and blood chemistry), vitals signs (hr and bp), physical examination. | up to 48 weeks

SECONDARY OUTCOMES:
to assess whether prolonged use of aerosolized tobramycin is required to sustain FEV1 increase (FEV1 expressed in liters and % predicted) | up to 48 weeks
Categorical results of microbiological tests referred to P. aeruginosa (negativisation, persistence, superinfection, re-infection); susceptibility testing of isolated P. aeruginosa strains (MIC90 and MIC50) | up to 48 weeks
Changes in body weight and BMI | up to 48 weeks
to assess health related quality of life | Initial visit, Week 20, Week 44

CONTACTS AND LOCATIONS:
Overall Officials: Henryk Mazurek, Doctor, Principal Investigator — Klinika Pneumonologii i Mukowiscydozy, Instytut Gruzlicy i Chorob Pluc w Rabce Zdroj
Locations (20):
- France (3):
  - CHR Clemenceau, Caen
  - Hopital Arnaud de Villeneuve, Clinique des maladies respiratoires, Montpellier
  - Hopital Necker, Paris
- Poland (8):
  - Specjalistyczny ZOZ nad Matka i Dzieckiem, Poradnia Leczenia Mukowiscydozy, Gdansk
  - I Oddzial Chorob Dzieciecych, Wojewodzki Specjalistyczny Szpital Dzieciecy, Kielce
  - Oddzial Kliniczny Interny Dzieciecej i Alergologii, Wojewodzki Szpital Specjalistyczny, Lodz
  - Dzieciecy Szpital Kliniczny Akademii Medycznej, Klinika Chorob Pluc I Reumatologii, Lublin
  - Klinika Pneumonologii, Alergologii Dzieciecej i Immunologii Klinicznej Szpital Kliniczny Uniwersytetu Medycznego w Poznaniu, Poznan
  - Klinika Pneumonologii i Mukowiscydozy, Instytut Gruzlicy i Chorob Pluc w Rabce Zdroj, Rabka-Zdrój
  - Poradnia Mukowiscydozy Wojewodzkiej, Przychodni Specjalistycznej dla Dzieci, Szpitala Wojewodzkiego Nr 2, Rzeszów
  - Klinika Pediatrii Instytut Matki I Dziecka, Warsaw
- Ukraine (9):
  - Dnipropetrovsk City Children Clinical Hospital # 2, Dnipropetrovsk
  - Donetsk Regional Children Clinical Hospital, Donetsk
  - Kriviy Rig City Clinical Hospital # 8, Kryvyi Rih
  - Institute of Phthysiology and Pulmonology n.a., F.G.Yanovskiy of the Academy of Medical Science of Ukraine, Kyiv
  - Institute of Pediatrics, Obstetrics and Gynecology of the Academy of Medical Science of Ukraine, Kyiv
  - Lviv Regional Children Specialized Clinical Hospital, Lviv
  - Odesa Regional Children Clinical Hospital, Odesa
  - Simferopol Central District Clinical Hospital, Simferopol
  - Zaporizhya Regional Clinical Children Hospital, Zaporizhya

REFERENCES:
- [Background] Wine JJ. Cystic fibrosis: How do CFTR mutations cause cystic fibrosis? Curr Biol. 1995 Dec 1;5(12):1357-9. doi: 10.1016/s0960-9822(95)00269-7. No abstract available. PMID 8749384
- [Background] Lewis PA. The epidemiology of cystic fibrosis. In: Hodson ME, Geddes DM. Cystic Fibrosis 2nd edition, Arnold, London 2000; 1a: 2-12.
- [Background] Dodge JA, Morison S, Lewis PA, Coles EC, Geddes D, Russell G, Littlewood JM, Scott MT. Incidence, population, and survival of cystic fibrosis in the UK, 1968-95. UK Cystic Fibrosis Survey Management Committee. Arch Dis Child. 1997 Dec;77(6):493-6. doi: 10.1136/adc.77.6.493. PMID 9496181
- [Background] Lucotte G, Hazout S, De Braekeleer M. Complete map of cystic fibrosis mutation DF508 frequencies in Western Europe and correlation between mutation frequencies and incidence of disease. Hum Biol. 1995 Oct;67(5):797-803. PMID 8543293
- [Background] Bossi A, Battistini F, Braggion C, Magno EC, Cosimi A, de Candussio G, Gagliardini R, Giglio L, Giunta A, Grzincich GL, La Rosa M, Lombardo M, Lucidi V, Manca A, Mastella G, Moretti P, Padoan R, Pardo F, Quattrucci S, Raia V, Romano L, Salvatore D, Taccetti G, Zanda M. [Italian Cystic Fibrosis Registry: 10 years of activity]. Epidemiol Prev. 1999 Jan-Mar;23(1):5-16. Italian. PMID 10356860
- [Background] Yamashiro Y, Shimizu T, Oguchi S, Shioya T, Nagata S, Ohtsuka Y. The estimated incidence of cystic fibrosis in Japan. J Pediatr Gastroenterol Nutr. 1997 May;24(5):544-7. doi: 10.1097/00005176-199705000-00010. PMID 9161949
- [Background] Imaizumi Y. Incidence and mortality rates of cystic fibrosis in Japan, 1969-1992. Am J Med Genet. 1995 Aug 28;58(2):161-8. doi: 10.1002/ajmg.1320580215. PMID 8533810
- [Background] Boat TF, Welsh MJ, Beaudet AL. Cystic fibrosis, in the metabolic basis of inherited disease (7th edn). McGraw-Hill, New York,1995.
- [Background] Wood RE, Boat TF, Doershuk CF. Cystic fibrosis. Am Rev Respir Dis. 1976 Jun;113(6):833-78. doi: 10.1164/arrd.1976.113.6.833. No abstract available. PMID 779549
- [Background] Rommens JM, Iannuzzi MC, Kerem B, Drumm ML, Melmer G, Dean M, Rozmahel R, Cole JL, Kennedy D, Hidaka N, et al. Identification of the cystic fibrosis gene: chromosome walking and jumping. Science. 1989 Sep 8;245(4922):1059-65. doi: 10.1126/science.2772657.
- [Background] Riordan JR, Rommens JM, Kerem B, Alon N, Rozmahel R, Grzelczak Z, Zielenski J, Lok S, Plavsic N, Chou JL, et al. Identification of the cystic fibrosis gene: cloning and characterization of complementary DNA. Science. 1989 Sep 8;245(4922):1066-73. doi: 10.1126/science.2475911.
- [Background] Anderson MP, Gregory RJ, Thompson S, Souza DW, Paul S, Mulligan RC, Smith AE, Welsh MJ. Demonstration that CFTR is a chloride channel by alteration of its anion selectivity. Science. 1991 Jul 12;253(5016):202-5. doi: 10.1126/science.1712984.
- [Background] Trapnell BC, Chu CS, Paakko PK, Banks TC, Yoshimura K, Ferrans VJ, Chernick MS, Crystal RG. Expression of the cystic fibrosis transmembrane conductance regulator gene in the respiratory tract of normal individuals and individuals with cystic fibrosis. Proc Natl Acad Sci U S A. 1991 Aug 1;88(15):6565-9. doi: 10.1073/pnas.88.15.6565. PMID 1713683
- [Background] Høiby N. Microbiology of lung infections in cystic fibrosis patients. Acta Paediatr Scand 1982; 301: 33-54.
- [Background] Moss RB, Babin S, Hsu YP, Blessing-Moore J, Lewiston NJ. Allergy to semisynthetic penicillins in cystic fibrosis. J Pediatr. 1984 Mar;104(3):460-6. doi: 10.1016/s0022-3476(84)81117-8. PMID 6323664
- [Background] Hodson ME, Gallagher CG, Govan JR. A randomised clinical trial of nebulised tobramycin or colistin in cystic fibrosis. Eur Respir J. 2002 Sep;20(3):658-64. doi: 10.1183/09031936.02.00248102. PMID 12358344
- [Background] Ramsey BW, Dorkin HL, Eisenberg JD, Gibson RL, Harwood IR, Kravitz RM, Schidlow DV, Wilmott RW, Astley SJ, McBurnie MA, et al. Efficacy of aerosolized tobramycin in patients with cystic fibrosis. N Engl J Med. 1993 Jun 17;328(24):1740-6. doi: 10.1056/NEJM199306173282403. PMID 8497284
- [Background] Ramsey BW, Pepe MS, Quan JM, Otto KL, Montgomery AB, Williams-Warren J, Vasiljev-K M, Borowitz D, Bowman CM, Marshall BC, Marshall S, Smith AL. Intermittent administration of inhaled tobramycin in patients with cystic fibrosis. Cystic Fibrosis Inhaled Tobramycin Study Group. N Engl J Med. 1999 Jan 7;340(1):23-30. doi: 10.1056/NEJM199901073400104. PMID 9878641
- [Background] Gilligan PH. Microbiology of airway disease in patients with cystic fibrosis. Clin Microbiol Rev. 1991 Jan;4(1):35-51. doi: 10.1128/CMR.4.1.35. PMID 1900735
- [Background] Ramsey BW, Schaeffler BL, Montgomery AB, et al. Survival and lung function during two years of treatment with intermittent tobramycin solution for inhalation in CF patients. Presented at European Cystic Fibrosis Conference (June 1999), The Hague, The Netherlands.
- [Background] Van Dalfsen JM, Lin L, Burns JL, et al. Microbiology effect of 18 months of intermittent inhaled tobramycin in patients with CF. Presented at European Cystic Fibrosis Conference (June 1999), The Hague, The Netherlands.
- [Background] Lenoir G, Aryayev N, et al. Highly concentrated aerosolized Tobramycin in the treatment of patients with cystic fibrosis and Pseudomonas aeruginosa infection. Eur. Respir. J 2005:26 (suppl. 49) 620s.
- [Background] Chuchalin A, Gyurkovics K, et al. Long term administration of aerosolised tobramycin, in patients with cystic fibrosis. Eur. Respir. J.2005: 26 (suppl 49) 3942s.
- [Background] Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung volumes and forced ventilatory flows. Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl. 1993 Mar;16:5-40. No abstract available. PMID 8499054
- [Background] Pin I, Gibson PG, Kolendowicz R, Girgis-Gabardo A, Denburg JA, Hargreave FE, Dolovich J. Use of induced sputum cell counts to investigate airway inflammation in asthma. Thorax. 1992 Jan;47(1):25-9. doi: 10.1136/thx.47.1.25. PMID 1539140
- [Background] Henry DA, Campbell ME, LiPuma JJ, Speert DP. Identification of Burkholderia cepacia isolates from patients with cystic fibrosis and use of a simple new selective medium. J Clin Microbiol. 1997 Mar;35(3):614-9. doi: 10.1128/jcm.35.3.614-619.1997. PMID 9041399
- [Background] Bauernfeind A, Rotter K, Weisslein-Pfister C. Selective procedure to isolate haemophilus influenzae from sputa with large quantities of Pseudomonas aeruginosa. Infection. 1987 Jul-Aug;15(4):278-80. doi: 10.1007/BF01644138. PMID 3117701
- [Background] Johansen HK, Hoiby N. Seasonal onset of initial colonisation and chronic infection with Pseudomonas aeruginosa in patients with cystic fibrosis in Denmark. Thorax. 1992 Feb;47(2):109-11. doi: 10.1136/thx.47.2.109. PMID 1549817
- [Result] Mazurek H, Chiron R, Kucerova T, Geidel C, Bolbas K, Chuchalin A, Blanco-Aparicio M, Santoro D, Varoli G, Zibellini M, Cicirello HG, Antipkin YG. Long-term efficacy and safety of aerosolized tobramycin 300 mg/4 ml in cystic fibrosis. Pediatr Pulmonol. 2014 Nov;49(11):1076-89. doi: 10.1002/ppul.22989. Epub 2014 Jan 24. PMID 24464974
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=CMA-0631-PR-0010